CLINICAL TRIAL: NCT04699383
Title: Documentation of Patient Outcomes for the Combination Treatment of Sodium Stibogluconate and Allopurinol in Complicated Cutaneous Leishmaniasis in Ethiopia
Brief Title: Documentation of Patient Outcomes for SSG/Allopurinol Combination Treatment in Ethiopia
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Wollo University (Other); Boru Meda Hospital (Unknown); University of Gondar (Other)
Responsible Party: Sponsor
Other Study IDs: 1361/20
Record Dates: First submitted 2020-10-19; First posted 2021-01-07 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Cutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Antimony Sodium Gluconate; Allopurinol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 3mm Punch biopsy at baseline (optional), 4mL serum and 4 non-invasive tape sampling discs at every study visit (optional).
  Storage of routinely taken Giemsa-stained microscopy slide of skin slit smear sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Sodium Stibogluconate with allopurinol — Routine administration of SSG/allopurinol combination treatment, from 1-5 cycles

SUMMARY:
Outcomes of patients receiving SSG and Allopurinol combination have never been documented systematically in Ethiopia. Therefore, it is not known how effective this combination is. This study will provide evidence to help clinicians make the best choice regarding treatment for complicated cutaneous leishmaniasis (CL) cases. Due to diversity in host-pathogen interactions across the different CL forms, early immunological correlates associated with treatment responsiveness and unresponsiveness could help treatment recommendation and provide us with the basis to develop new diagnostic and treatment strategies.

This study aims to document treatment outcomes of patients with cLCL, MCL, and DCL receiving systemic treatment using SSG and Allopurinol combination within a routine care setting located in a highly endemic area in Ethiopia.

DETAILED DESCRIPTION:
Cutaneous Leishmaniasis (CL) in Ethiopia causes severe dermatological mutilations. Forms that require systemic treatment are complicated localized cutaneous leishmaniasis (cLCL), mucocutaneous leishmaniasis (MCL), and diffuse cutaneous leishmaniasis (DCL). The clinical presentation of CL depends on various factors including parasite species, infection history and differences in the immune response. National guidelines recommend equally all drugs that are also used for visceral leishmaniasis treatment. Sodium stibogluconate (SSG) is one of these recommended medications. However, dermatologists in Ethiopia also use a combination of SSG and Allopurinol for treatment of complicated cutaneous leishmaniasis.

Outcomes of patients receiving SSG and Allopurinol combination have never been documented systematically in Ethiopia. Therefore, it is not known how effective this combination is. This study will provide evidence to help clinicians make the best choice regarding treatment for complicated CL cases. Due to diversity in host-pathogen interactions across the different CL forms, early immunological correlates associated with treatment responsiveness and unresponsiveness could help treatment recommendation and provide us with the basis to develop new diagnostic and treatment strategies.

This study aims to document treatment outcomes of patients with cLCL, MCL, and DCL receiving systemic treatment using SSG and Allopurinol combination within a routine care setting located in a highly endemic area in Ethiopia.

ELIGIBILITY:
Inclusion Criteria:

* Clinically or microscopically confirmed diagnosis of MCL, DCL or complicated LCL
* Clinical routine care decision to initiate systemic CL treatment using SSG with allopurinol
* Willing and able to provide informed consent

Exclusion Criteria:

* Medical emergencies, underlying chronic conditions or other circumstances that make participation in this study medically or otherwise inadvisable

Study sample collection only for Age 18 and above

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cLCL, MCL, or DCL who present during the study period, either referred from peripheral facilities or self-referred, and who receive systemic CL treatment using SSG and allopurinol will be invited to be included in the study consecutively. The decision whether or not to use SSG and Allopurinol in a patient is part of routine care.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Treatment outcome at day 180 (proportion with cure, good response, poor response, no response and relapse) | day 180
  cure defined as 100% flattening and/or reepithelization, good response 50-99% flattening and/or reepithelization, poor response 1-49% flattening and/or reepithelization, no response 0% flattening and/or reepithelization and relapse as worsening of existing lesion or appearance of new lesions

SECONDARY OUTCOMES:
Patient reported outcomes using the dermatology life quality index (DLQI) | day 0 - day 180
  Mean difference in Dermatology life quality index (min 0, max 30) before treatment and at day 180
Side-effects | day 0 - day 180
  Proportion of patients with side-effects and proportion of side-effects according to CTCAE severity grades
Cycles to cure | day 0 - day 180
  Number of cycles needed to reach cure
Factors associated with cure | day 30, day 180
  To determine covariate-adjusted risk ratios for baseline and follow-up factors associated with cure after one cycle of treatment and at the end of cycle 5
Treatment outcome at day 30 (proportion with cure, good response, poor response, and no response ) | day 30
  cure defined as 100% flattening and/or reepithelization, good response 50-99% flattening and/or reepithelization, poor response 1-49% flattening and/or reepithelization, no response 0% flattening and/or reepithelization

CONTACTS AND LOCATIONS:
Locations (1):
- Boru Meda Hospital, Dessie, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Henten S, Bialfew F, Hassen S, Tilahun F, van Griensven J, Abdela SG. Treatment of Cutaneous Leishmaniasis with Sodium Stibogluconate and Allopurinol in a Routine Setting in Ethiopia: Clinical and Patient-Reported Outcomes and Operational Challenges. Trop Med Infect Dis. 2023 Aug 14;8(8):414. doi: 10.3390/tropicalmed8080414. PMID 37624352